CLINICAL TRIAL: NCT00249860
Title: A Multicentre Phase III Study of Interferon-beta-1a for the Treatment of Chronic Hepatitis C in Asian Subjects
Brief Title: A Multicenter Phase 3 Study of Interferon-beta-1a for the Treatment of Chronic Hepatitis C in Asian Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck Pte. Ltd., Singapore (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23744
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C
Keywords: Subjects with chronic hepatitis C who have never previously received interferon therapy.
MeSH Terms: conditions — Hepatitis C | interventions — Interferon beta-1a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Interferon-beta-1a (Experimental)
  Interventions: Drug: Interferon-beta-1a
- Ribavarin plus interferon-beta-1a (Active Comparator)
  Interventions: Drug: Placebo; Drug: Ribavirin plus Interferon-beta-1a

INTERVENTIONS:
Drug: Interferon-beta-1a — Interferon-beta-1a will be administered subcutaneously at a dose of 44 microgram (mcg), three times a week up to Week 24
  Arms: Interferon-beta-1a
Drug: Placebo — Matching placebo will be administered subcutaneously three times a week for 12 weeks. The placebo responders will continue the study off-treatment after Week 12 up to Week 24
  Arms: Ribavarin plus interferon-beta-1a
Drug: Ribavirin plus Interferon-beta-1a — Placebo non-responders at Week 12 will receive ribavirin at a dose of 1000 milligram (mg) or 1200 mg orally once daily in combination with Interferon-beta-1a, administered subcutaneously at a dose of 44 mcg three times a week, from Week 16 up to Week 24
  Arms: Ribavarin plus interferon-beta-1a

SUMMARY:
The main objective of this study is to establish interferon-beta-1a as the treatment of choice for chronic Hepatitis C with better efficacy and safety profiles in monotherapy or combination therapy.

This will be a multicenter, randomized, double-blind, placebo-controlled study with a placebo to be crossed-over to a combination of interferon-beta-1a and ribavirin or no treatment during an open-label extension phase. The duration of the trial will be 48 weeks, with a double-blind period of 12 weeks.

The study will recruit 257 eligible subjects of either sex. It will be conducted by approximately 16 Investigators / investigational centers in 3 countries (China, Hong Kong and Singapore).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Have an elevated serum alanine aminotransferase (ALT) between 1.5 and 10 times the upper limit of normal
* Had adequate bone marrow reserve and organ function
* Are not pregnant and are willing to use contraception, if, of childbearing potential
* Are willing and able to comply with the protocol and to give written informed consent
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Clinical evidence of liver cirrhosis or a diagnosis of definite cirrhosis on liver biopsy
* History of liver failure, severe retinopathy, immunologically mediated disease, cancer or epilepsy with a history of inadequately controlled seizures
* Any cause for the liver disease other than chronic hepatitis C
* Evidence of chronic renal impairment, liver cancer, unstable psychiatric disorder, known or ongoing alcohol or drug abuse
* Positive test at screening for Hepatitis B surface antigen, immunoglobulin M Hepatitis B core antibody and human immunodeficiency virus antibody
* Previous systemic treatment for Hepatitis C with an interferon or ribavirin
* Presence of systemic disease that might interfere with subject safety, compliance or evaluation
* Known allergies to acetaminophen, human serum albumin or mannitol;
* Glucocorticosteroids or other immunosuppressive drugs taken within 28 days of starting treatment
* Bearing organ transplants (except cornea)
* Other protocol defined exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2002-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving sustained viral response (SVR) at Week 24 | Week 24
Percentage of subjects achieving sustained viral response (SVR) at Week 48 | Week 48

SECONDARY OUTCOMES:
Change from baseline in viral load (Hepatitis C virus ribonucleic acid [HCV RNA]) at Week 12, 24, and 48 | Baseline, Week 12, 24, and 48
Percentage of subjects with Alanine transaminase (ALT) normalization | Week 12, 24, and 48
Percentage of subjects with viral clearance | Week 12 and 24
Percentage of subjects with both SVR and sustained ALT normalization | Week 48
Number of subjects with improvement in the liver necroinflammation score by at least two points | Week 48
Number of subjects with improvement in architectural staging (liver fibrosis) by at least one point | Week 48
Number of subjects with adverse events and serious adverse events | Baseline up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Wee, M.D., Study Director — Serono Singapore Ltd, an affiliate of Merck Serono SA, Singapore

REFERENCES:
- [Result] Chan HL, Ren H, Chow WC, Wee T; Interferon beta-1a Hepatitis C Study Group. Randomized trial of interferon beta-1a with or without ribavirin in Asian patients with chronic hepatitis C. Hepatology. 2007 Aug;46(2):315-23. doi: 10.1002/hep.21683. PMID 17654600
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com